CLINICAL TRIAL: NCT02734836
Title: Drug Eluting Stent for the Management of PERipheraal Arterial Disease of the SFA (DESPERADO-SFA Study)
Brief Title: Drug Eluting Stent for the Management of PERipheral Arterial Disease Of the SFA (DESPERADO-SFA Study)
Acronym: DESPERADO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AHH-2016-020
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty, Balloon; Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zilver PTX Stent (Experimental): Diagnostic assessment of the lesion after implantation of drug eluting stent with Balloon Angioplasty and placement of the Zilver PTX Stent with Optical Coherence Tomography (OCT)
  Interventions: Device: Balloon Angioplasty; Other: Optical Coherence Tomography

INTERVENTIONS:
Device: Balloon Angioplasty
Other: Optical Coherence Tomography

SUMMARY:
This is a prospective, nonrandomized, single-arm study using the Zilver PTXTM stent in patients with Superficial Femoral Artery (SFA) disease (total occlusions or significant stenosis).

DETAILED DESCRIPTION:
Endovascular therapy is widely used for the treatment of peripheral artery disease (PAD). Primary nitinol stenting for superficial femoral artery (SFA)) lesions has been shown to be superior to balloon angioplasty alone. Zilver PTX a paclitaxel -eluting nitinol stent has been approved by the Food and Drug Administration (FDA) for femoro-popliteal artery use. Previous study have reported safety and effectiveness of the Zilver PTZ in patients with de novo or re-stenotic lesions of the femoro-popliteal artery.

Optical Coherence tomography (OCT) is a novel intravascular imaging modality with a unique and fine resolution of 10 µm at the level of a red blood cells providing detailed images of vascular wall following stent implantation for evaluation of optimal stent apposition and expansion as well as intraluminal clot.

20 patients with symptomatic critical limb ischemia (CLI) and claudication without CLI (Rutherford class 2-6) and identifiable SFA disease on angiogram requiring percutaneous peripheral intervention (PPI)will be enrolled in this study. We would like to study the vessel apposition and expansion immediately after initial implantation as well as evaluation of late stent malapposition and neointimal hyperplasia at the 12 months follow up after Zilver PTXTM stent implantation using intravascular OCT imaging. Follow up visits will take place at 1 month, 6 month, 12 month and 13 month after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient with lower extremity claudication and Peripheral Arterial Disease (PAD) due to significant SFA stenosis (60%≤99%) or total occlusions (100%) that affects the quality of life despite medical therapy.
* Evidence of significant SFA disease involving the most symptomatic limb by noninvasive vascular testing with the use of the following:

  * ABI: <0.9 (If ABI>1.4, SFA systolic acceleration time should be > 140 milliseconds);
  * TBI: <0.6;
  * Computed Tomographic Angiography (CTA) confirming at least a 60% SFA stenosis; or
  * Magnetic Resonance Angiography (MRA) confirming at least a 60% SFA stenosis
* At least one patent, non-treated below the knee vessel.
* Male and female patients that are ≥ 18 years of age.
* Subject has been advised of the beneficial effects of smoking cessation and regular exercise but must not be in the process of changing their smoking status at the time of screening. Patients may resume or increase exercising as an effect of post procedurally improved lower limb perfusion.
* Peak Walking Time (PWT) limited only by claudication.
* Willingness to participate in the study, documented by signed, written informed consent.

Exclusion Criteria:

* Planned usage of atherectomy devices during procedure. The following devices are the only permitted devices that can be used for intervention procedures:

  * Conventional balloons
  * Zilver PTXTM stent
* Planned amputation.
* Any planned/scheduled revascularization procedures ≤ 30 days after baseline procedure.
* Prior lower extremity revascularization ≤ 30 days before baseline procedure.
* The target lesion is an in-stent restenosis.
* Infra-popliteal disease involving the last remaining vessel.
* Patients with a creatinine clearance < 30mL/min.
* Patients with known bleeding disorders.
* Patients with known active pathological bleeding.
* Patients with known hypersensitivity to acetylsalicylic acid, clopidogrel bisulfate, ticagrelor, Aspirin, or other antiplatelets/anticoagulants.
* Patients with known history of intracranial hemorrhage at any time, GI bleed in the past 6 months, or major surgery within the past 30 days.
* Patients with known ischemic stroke during the past 3 months.
* Patients with known severe liver disease.
* Patient with known history of congestive heart failure (CHF) with an LVEF of < 30%.
* Patients considered being at risk of bradycardic events unless treated with a permanent pacemaker.
* Female patients with known pregnancy, breast feeding, or intend to become pregnant during the study period (all female patients 55 years and younger, without a history of hysterectomy must have a pregnancy test prior to PPI at baseline and at 12 months).
* Concern for inability of the patient to comply with study procedures and/or follow up (e.g., alcohol or drug abuse).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Optimal Coherence Tomograpy | 12 Month
  Identification of optimal stent apposition and expansion as well as identification of intraluminal clot at 12 month post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Cilingiroglu, MD, Principal Investigator — Arkansas Heart Hospital; Gerardo Rodriguez, MD PhD, Study Director — Arkansas Heart Hospital
Locations (1):
- Arkansas Heart Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No